CLINICAL TRIAL: NCT04645628
Title: Optimization of the Acquisition Sequence to Improve the Quality and Comfort of Magnetic Resonance Imaging Exam
Acronym: AIMANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Valérie LAURENT, MD, PhD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A01969-30
Record Dates: First submitted 2020-11-16; First posted 2020-11-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects; Patient Performing an MRI Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects will have an MRI examination (Experimental)
  Interventions: Other: MRI examination

INTERVENTIONS:
Other: MRI examination — All subjects (healthy subjects and patients) will have an MRI examination with optimized sequences

SUMMARY:
The purpose of this study is to evaluate the optimization of MRI acquisition sequences.

ELIGIBILITY:
Inclusion Criteria for all subjects :

* to be over 18 year-old,
* to be able to understand the instructions given,
* to be enrolled in a social security plan,
* to have underwent a pre-inclusion medical examination,
* to give a written consent.

Inclusion Criteria especially for Patients :

* to perform a MRI examination of the head, neck, spine, thorax, abdomen, pelvis, retroperitoneum, lower limbs, upper limbs or whole body during clinical follow-up care.

Exclusion Criteria for all subjects :

* any contraindication to MR examination (active medical device, ferromagnetic foreign body, pregnancy, morbid obesity, claustrophobia, … ),
* subject under a measure of legal protection.

Exclusion Criteria especially for Healthy Subjects :

* to have a pathology in the anatomical area to be imaged
* to be employed by the CHRU of Nancy or having the slightest link of subordination with the CHRU of Nancy.

Exclusion Criteria especially for Patients :

* to have a limited MRI examination time due to a sensitive clinical situation (sedation, unstable hemodynamic state, postoperative).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2027-12-08 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Image quality based on standard imaging quality criteria. | 6 months after the last inclusion
  The image quality will be appreciated visually at least by a radiologist or a researcher.

SECONDARY OUTCOMES:
Comparison of the Signal to Noise Ratio obtained by the optimized MRI sequence and the reference situation (standard sequence). | 6 months after the last inclusion
  Signal to Noise Ratio will be measured in arbitrary units.
Comparison of the Contrast to Noise Ratio obtained by the optimized MRI sequence and the reference situation (standard sequence). | 6 months after the last inclusion
  Contrast to Noise Ratio will be measured in arbitrary units.
Comparison of the acquisition time obtained with the optimized MRI sequence and the reference situation (standard sequence). | 6 months after the last inclusion
  Time acquisition will be evaluated in minutes.
Comparison of blurring and artefacts obtained by the optimized MRI sequence and the reference situation (standard sequence). | 6 months after the last inclusion
  Absence of blurring and artefacts will be assessed by at least one radiologist according to an ordinal scale.
Comparison of the spatial resolution obtained by the optimized MRI sequence and the reference situation (standard sequence). | 6 months after the last inclusion
  Spatial resolution will be measured in mm².
Qualification of the MRI acquisition for a clinical study. | 6 months after the inclusion
  Validation of MRI acquisition by a centralized review center.
Evaluation of intra-subject reproducibility on the same MRI and on two MRIs. | 6 months after the last inclusion
  Measurement of intra-subject reproducibility on the same MRI and on two MRIs by the intra-class correlation coefficient for quantitative measurement or by the kappa coefficient for a qualitative measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France